CLINICAL TRIAL: NCT02277184
Title: A Phase 1b Study of Ficlatuzumab, Cisplatin and Intensity Modulated Radiotherapy (IMRT) in Intermediate or High Risk, Previously Untreated, Locally Advanced Head and Neck Squamous Cell Carcinoma With Biomarker Correlatives
Brief Title: Ficlatuzumab, Cisplatin and IMRT in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the investigator left the institution
Sponsor: Julie E. Bauman, MD, MPH (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Julie E. Bauman, MD, MPH, Director of the Head and Neck Cancer Section and Thyroid Cancer Section in the Division of Hematology-Oncology at the University of Pittsburgh School of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-060
Record Dates: First submitted 2014-10-25; First posted 2014-10-28 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: Intermediate Risk HNSCC; High Risk HNSCC; Previously Untreated, Locally Advanced HNSCC; Undifferentiated carcinoma; Poorly differentiated carcinoma of the oral cavity; Poorly differentiated carcinoma of the oropharynx; Poorly differentiated carcinoma of the larynx; Poorly differentiated carcinoma of the hypopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma | interventions — ficlatuzumab; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ficlatuzumab, Cisplatin and IMRT (Experimental): Ficlatuzumab will be administered as an IV infusion over 30-60 minutes, once every two weeks beginning the week prior to cisplatin-IMRT (week -1), for a total of 4 doses.
  Cisplatin will be administered as an IV infusion over 60 minutes on Monday, Tuesday, or Wednesday of each treatment week beginning concurrent with IMRT during week 1 of study treatment (and one week following the first dose of ficlatuzumab) for a total of 7 doses.
  IMRT: Treatment will be delivered once daily, 5 fractions per week, 35 - 37 fractions, no weekends or holidays over 7 - 8 weeks. All targets will be treated sequentially.
  Interventions: Drug: Ficlatuzumab; Drug: Cisplatin; Radiation: Intensity Modulated Radiotherapy (IMRT)

INTERVENTIONS:
Drug: Ficlatuzumab — Ficlatuzumab Concentrate for Injection, 20 mg/mL, is formulated in 10 mM histidine buffer pH 5.8. The formulation also includes 142 mM arginine (for isotonicity) and 0.01% polysorbate 80. The product is sterile filtered and aseptically filled into washed and depyrogenated 5 mL glass vials.The product is a clear to slightly opalescent, colorless to slightly yellow, solution.
  Ficlatuzumab Concentrate for Injection is to be administered by IV infusion as an admixture with normal saline solution. The admixture solution in an IV bag is connected to an infusion set containing a 0.22 µm low protein-binding in line filter. The filtered admixture solution is clear to slightly opalescent.
  Ficlatuzumab is to be stored under refrigerated conditions (2C - 8C)
  Other Names: AV-299; SCH900 105
Drug: Cisplatin — Each vial contains 10 mg of DDP, 19 mg of sodium chloride, 100 mg of mannitol, and hydrochloric acid for pH adjustment. One vial is reconstituted with 10 ml of sterile water. The pH range will be 3.5 to 4.5.
  Cisplatin will be given as a bolus, infused over 1-2 hours along with appropriate hydration and anti-emetics.
  Reconstituted solution of cisplatin is stable for 20 hours when stored at 27°C and should be protected from light if not used within 6 hours. The vials and injection should not be refrigerated. Cisplatin has been shown to react with aluminum needles, producing a black precipitate within 30 minutes.
  Other Names: PLATINOL
Radiation: Intensity Modulated Radiotherapy (IMRT) — Immobilization should be performed to ensure daily reproducibility of setup.Treatment planning CT scans will be required to define tumor, clinical and planning target volumes.The treatment planning CT scan should be performed with IV contrast. All tissues to be irradiated must be included in the CT scan.
  Targets are defined as primary (requiring a higher dose) and secondary (targets at lower risk requiring a lower dose). The primary target is the PTV3 of the primary tumor and lymph nodes containing clinical or radiographic evidence of metastases. The secondary target is the PTVs consist of an area at intermediate risk (PTV2) and that containing the lowest risk of lymph node involvement (PTV2).
  The treatment plan will be based on an analysis of the volumetric dose, including dose volume histogram (DVH) analyses of the PTV and critical normal structures. Inverse planning will be utilized to deliver optimal dose to the PTVs while excluding noninvolved normal tissue.

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is the most common cancer arising in the upper aerodigestive tract, and is the sixth leading incident cancer worldwide. Despite advances in multimodality therapy, 5-year overall survival (OS) is 40-60%, and has increased only incrementally in the past two decades. The current standard of care for primary nonsurgical management of locally advanced HNSCC is concurrent cisplatin-radiotheray, which significantly improved OS, progression-free survival, and locoregional control compared with radiotherapy alone in the landmark Intergroup trial 0126.

The MET proto-oncogene encodes c-Met, a heterodimeric growth factor receptor bound exclusively by its ligand, hepatocyte growth factor (HGF). In the laboratory, activation of the HGF/c-Met pathway is associated with resistance to cisplatin and radiotherapy in HNSCC. We hypothesize that the addition of an HGF/c-Met pathway inhibitor to cisplatin-radiotherapy may improve outcomes in HNSCC. Ficlatuzumab (AV-299) is a humanized HGF-inhibitory IgG1 monoclonal antibody.

The primary objective of this study is to establish the recommended phase II dose (RP2D) of the combination of ficlatuzumab, cisplatin and intensity-modulated radiotherapy (IMRT), in patients with locally advanced HNSCC. The dose-finding study design will follow a Narayana k-in-a-row design with k set to 3 to target a 33% DLT rate. In the dose-finding phase, a total of either 10 or 14 patients will be treated. If no DLTs are observed among 10 patients, the highest dose tier will be declared the RP2D. Otherwise the RP2D will be estimated from DLTs across all dose levels by isotonic regression. The secondary objective is to estimate biomarker association with preliminary clinical response. We will evaluate biomarkers of HGF/cMet pathway activation in tumor tissue, plasma, and immune cells.

DETAILED DESCRIPTION:
This will be a phase Ib trial where ficlatuzumab will be added to the standard of care for locally advanced HNSCC: cisplatin-IMRT. Biomarkers of HGF/cMet pathway activation that may associate with clinical response will be developed in an expansion cohort. Patients with high or intermediate risk, locally advanced HNSCC will be eligible.

A diagnostic primary tumor block for biomarker correlatives is mandatory for inclusion to this study. A representative paraffin block of the original diagnosis and all repeat biopsies, if available, will be submitted.

The starting dose of ficlatuzumab (dose tier 1) will be 10 mg/kg every 2 weeks, beginning the week prior to cisplatin-IMRT (week -1). Ficlatuzumab will be administered as an IV infusion over 30-60 minutes, for a total of 4 doses.

The starting dose of cisplatin (dose tier 1) will be 40 mg/m2 weekly, beginning concurrent with IMRT during week 1 of study treatment (and one week following the first dose of ficlatuzumab which is administered during week -1 of study treatment). Patients will receive cisplatin once weekly as an IV infusion over 60 minutes, for a total of 7 doses.

Megavoltage energy photon beam irradiation is required. Any treatment planning and delivery system that has been credentialed for head and neck IMRT is acceptable. Immobilization should be performed with a thermoplastic mask to ensure daily reproducibility of setup. Treatment planning CT scans will be required to define tumor, clinical and planning target volumes.The treatment planning CT scan should be acquired with the patient in the same position and immobilization device as for treatment and performed with IV contrast so that major vessels of the neck are easily visualized.

Four dose tiers will be considered for the phase I portion for ficlatuzumab and cisplatin. IMRT will remain consistent for all dose tiers. Under this schema, more than one patient can be enrolled at the same time. However de novo dose escalation cannot occur until 2 patients have completed study treatment without DLT. In the dose-finding phase, a total of 10 patients will be treated if no DLTs are observed or 14 patients if at least one DLT occurs. If no DLTs are observed among the first 10 patients the recommended for phase 2 dose (RP2D) will be set to dose tier 3. If a DLT is observed and 14 patients are treated and observed, the RP2D will be estimated from DLTs across all dose levels by isotonic regression. The observation period for identifying a DLT will be 10 weeks, or 2 weeks following completion of IMRT, whichever comes later. To be considered a DLT, the toxicity must be at least possibly related to ficlatuzumab. An expansion cohort will then proceed at RP2D until 12 patients have been treated at that dose level.

In the absence of treatment delays due to adverse event(s), treatment may continue until one of the following criteria applies:

* Completion of treatment,
* Disease progression,
* Intercurrent illness that prevents further administration of treatment,
* Unacceptable adverse event(s),
* Patient decides to withdraw from the study, or
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

After completing treatment, patients will be followed every 3 months for 2 years, then every 6 months for 3 years, for a total of 5 years from completion of IMRT. Patients removed from study for unacceptable adverse event(s) will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Patients must have histologically confirmed squamous cell carcinoma, undifferentiated carcinoma, or poorly differentiated carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx with no evidence of distant metastasis. Biopsy sampling of primary tumor with pathology report documentation of confirmed diagnostic tissue type is required. Patients should be evaluated by a Radiation Oncologist, Medical Oncologist and Otolaryngologist prior to enrolling on study.
* Patients must have high risk or intermediate risk disease, defined below. Staging evaluation should be determined by imaging studies and complete head and neck exam in accordance with the American Joint committee on Cancer Staging Manual, 7th edition

  o High risk patients must meet one of the following criteria:
* Unresectable oral cavity
* Larynx: T4 any N; T2-3 and ≥N2a
* Hypopharynx and p16(-) oropharynx: Stage III-IVb except T1N1
* p16(-) Oropharnyx: Stage III-IVb except T1N1

  o Intermediate risk, p16(+) oropharynx patients must meet one of the following criteria:
* T3 or ≥ N2a AND ≥10 pack-years tobacco exposure (See Tobacco Assessment Form, Appendix A)
* T4 disease, irrespective of smoking status
* N3 disease, irrespective of smoking status

Note: for oropharyngeal patients, p16 status must be known, and can be performed at the local site. p16-positive disease is defined as ≥70% of tumor cells demonstrating diffuse nuclear and cytoplasmic staining by p16 immunohistochemistry (IHC). A positive test for HPV-16 by in-situ hybridization (ISH), if this is the local site preference for assessing HPV status, may substitute for p16 IHC testing. p16 staining is not required for non-oropharyngeal sites.

* Patients must be untreated with curative-intent surgery for current diagnosis of Stage III, IVa, or IVb disease. Diagnostic biopsy of primary tumor and/or nodal sites is permitted.

  * Diagnostic simple tonsillectomy is permitted, provided patient has RECIST-measurable nodal disease.
  * Patients with a second HNSCC primary tumor are eligible for this study, provided more than 2 years have elapsed since the first diagnosis of HNSCC, the original tumor was managed with surgery only (no adjuvant chemotherapy or radiotherapy), and has not recurred.
* Patients with simultaneous primaries or bilateral tumors are excluded, with the exception of patients with bilateral tonsil cancers or patients with T1-2, N0, M0 resected differentiated thyroid carcinoma, who are eligible.
* No prior systemic (chemotherapy or biologic/molecular targeted therapy) or radiation treatment for head and neck cancer.

  * Patients may have received chemotherapy or radiation for a previous, curatively treated non-HNSCC malignancy, provided at least 2 years have elapsed.
  * Patients must be untreated with radiation above the clavicles.
* Patients with a history of curatively-treated non-HNSCC malignancy must be disease-free for at least 2 years except for excised and cured: carcinoma-in-situ of breast or cervix; non-melanomatous skin cancer; T1-2, N0, M0 resected differentiated thyroid carcinoma; superficial bladder cancer; T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection.
* Diagnostic primary tumor tissue must be available for biomarker correlatives, in both the dose-finding and expansion cohorts.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 (See Appendix B)
* Age ≥ 18
* Patients must have measurable disease according to RECIST 1.1 (See Section 6.1)
* Patients must have the following laboratory values measured within 28 days of registration:

  * Absolute neutrophil count (ANC) > 1500/mm3
  * Hemoglobin (Hb) > 8.0 g/dL
  * Platelet count (PLT) > 100,000/mm3
  * Creatinine clearance ≥ 45 ml/min determined by 24-hour collection or estimated by the Cockraft-Gault formula:
  * Calculated Creatinine Clearance = [(140-age) X (actual body weight in kg) X (0.85 if female)]/(72 X serum creatinine)
  * Serum bilirubin < 2 mg/dL
  * AST (aspartate aminotransferase) and ALT (alanine aminotransferase) < 3 times upper limit of normal (ULN)
* No prior severe infusion reaction to a monoclonal antibody
* Written informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* If a woman of childbearing potential, documentation of negative pregnancy within 14 days prior to first dose. Sexually active patients must agree to use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug. All fertile female subjects (and their partners) must agree to use a highly effective method of contraception. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). Should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent.
* Distant metastatic disease including CNS or leptomeningeal metastases is not allowed.
* Left ventricular ejection fraction (LVEF) ≤ 50%.
* Significant pulmonary disease, including pulmonary hypertension or interstitial pneumonitis.
* Decreased serum albumin < 30 g/L (< 3 g/dL).
* Peripheral edema ≥ Grade 2 per NCI-CTCAE version 4.0.
* Significant electrolyte imbalance prior to enrollment:

  * Hypomagnesemia < 1.2 mg/dL or 0.5 mmol/L.
  * Hypocalcemia < 8.0 mg/dL or 2.0 mmol/L.
  * Hypokalemia < 3.0 mmol/L.
* Significant dermatological disease including but not limited to, skin drying and fissuring, paronychial inflammation, infectious sequelae (eg. blepharitis, cheilitis, cellulitis, cyst).
* Peripheral neuropathy ≥ Grade 2
* Significant cardiovascular disease, including:

  * Cardiac failure New York Heart Association (NYHA) class III or IV.
  * Myocardial infarction, severe or unstable angina within 6 months prior to Study Day 1.
  * History of serious arrhythmia (i.e., ventricular tachycardia, or ventricular fibrillation).
  * Cardiac arrhythmias requiring anti-arrhythmic medications.
* Significant thrombotic or embolic events within 3 months prior to Study Day 1. Significant thrombotic or embolic events include but are not limited to stroke or transient ischemic attack (TIA). Catheter-related thrombosis is not a cause for exclusion. Diagnosis of deep vein thrombosis or pulmonary embolism is allowed if it occurred > 3 months prior to Study Day 1 and the patient has completed or is on stable anti-coagulation therapy.
* Any other medical condition (eg, alcohol abuse) or psychiatric condition that, in the opinion of the Investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
* History of second malignancy within 2 years prior to Study Day 1 (except for excised and cured non-melanoma skin cancer, carcinoma in situ of breast or cervix, superficial bladder cancer, or T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection).
* Major surgery within 6 weeks prior to Study Day 1 (subjects must have completely recovered from any previous surgery prior to Study Day 1).
* Active infection requiring antibiotics or antifungals within 7 days prior to first dose of study drug.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with study drugs. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated. Note: HIV testing is not required for entry into this protocol.
* Women must not be pregnant or breastfeeding because chemotherapy and/or ficlatuzumab may be harmful to the fetus or the nursing infant. Pregnant women are excluded from this study because chemotherapy and/or ficlatuzumab have the potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Establish the recommended-for-phase II dose (RP2D) of the combination of ficlatuzumab, cisplatin and intensity-modulated radiotherapy (IMRT) | 1 year
  A dose escalation/de-escalation plan will be conducted according to an adaptive Narayana k-in-a-row design.We will select the dose of ficlatuzumab that is close to but does not exceed a 33% dose limiting toxicity (DLT) rate when administered with a fixed standard dose of cisplatin and IMRT. The observation period for identifying a DLT will be 10 weeks, or 2 weeks following completion of IMRT, whichever comes later. Note: to be considered a DLT, the toxicity must be at least possibly related to ficlatuzumab.In the dose-finding phase, a total of 10 patients will be treated if no DLTs are observed or 14 patients if at least one DLT occurs. If no DLTs are observed among the first 10 patients the recommended for phase 2 dose (RP2D) will be set to dose tier 3. If a DLT is observed and 14 patients are treated and observed, the RP2D will be estimated from DLTs across all dose levels by isotonic regression.

SECONDARY OUTCOMES:
Evaluate the preliminary efficacy of the combination of ficlatuzumab, cisplatin and intensity-modulated radiotherapy as curative-intent treatment for patients with locally advanced HNSCC | 5 years
  The preliminary clinical efficacy of the combination of ficlatuzumab, cisplatin and IMRT will be described according to CR rate (RECIST 1.1 and Integrated PET/CT criteria), median TTP, LRC, and median OS in: 1) the entire study population; 2) patients treated at RP2D.
  All patients will be evaluable for toxicity from the time of their first treatment with ficlatuzumab. The proportion of DLTs in each dosing cohort will be reported, as will the proportion of AEs in accordance with NCI CTCAE v.4 grading criteria
Evaluate biomarkers of HGF/c-Met pathway activation in baseline tumor biopsies, to correlate with preliminary efficacy data | 5 years
  Submission of primary tumor tissue for biomarker correlatives is mandatory to measure tumor protein levels of cMet and HGF prior to study treatment.
  The relationship of percent change in the baseline sum diameter of all measurable RECIST lesions to baseline cMet and HGF will be characterized by a linear, or if necessary, generalized linear or nonlinear regression model with appropriate confidence intervals.
Evaluate change in biomarkers of HGF/c-Met pathway activation after a single dose of ficlatuzumab, prior to initiation of cisplatin-IMRT, to correlate with preliminary efficacy data | 5 years
  Biomarkers in blood will be quantitatively measured and will be evaluated as predictors of tumor response in appropriate generalized linear models. Calculated p values for testing the significance of the prediction models will be adjusted for false discovery by the method of Benjamini and Hochberg.
Evaluate pharmacodynamic plasma biomarkers of HGF/c-Met pathway activation to correlate with preliminary efficacy data. | 5 years
  Biomarkers in blood will be quantitatively measured and will be evaluated as predictors of tumor response in appropriate generalized linear models. Calculated p values for testing the significance of the prediction models will be adjusted for false discovery by the method of Benjamini and Hochberg.
Describe the prevalence of PIK3CA, PTEN, and HRAS mutations in patients' tumors | 5 years
  The peripheral biomarkers related to HGF/c-Met pathway activation will be evaluated. Baseline values and changes in these biomarkers to quantitative response data and PFS will be evaluated. Biomarkers in tumor and blood will be quantitatively measured and will be evaluated as predictors of tumor response in appropriate generalized linear models. Calculated p values for testing the significance of the prediction models will be adjusted for false discovery by the method of Benjamini and Hochberg.
Describe dendritic and T cell phenotypes in pre and post ficlatuzumab biopsies | 5 years
  HNSCC is an immunosuppressive disease. Patients demonstrate lower absolute lymphocyte counts than healthy subjects, impaired natural killer (NK) cell activity and poor antigen-presenting function. Mechanistically, HGF inhibits dendritic cell activation. Evaluation of the dendritic cell and T cell phenotypes in baseline biopsies will be evaluated. In addition, longitudinal T cell and NK cell phenotypes in peripheral blood will be analyzed before, during and after exposure to ficlatuzumab.
Evaluate pharmacodynamic biomarkers of peripheral T cell and natural killer cell activation | 5 years
  HNSCC is an immunosuppressive disease. Patients demonstrate lower absolute lymphocyte counts than healthy subjects, impaired natural killer (NK) cell activity and poor antigen-presenting function. Mechanistically, HGF inhibits dendritic cell activation. Evaluation of the dendritic cell and T cell phenotypes in baseline biopsies will be evaluated. In addition, longitudinal T cell and NK cell phenotypes in peripheral blood will be analyzed before, during and after exposure to ficlatuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Bauman, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania